CLINICAL TRIAL: NCT00440219
Title: The Effect of Preoperative Oral Prednisone on the Operative Field During Nasal Polypectomy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, IWitterick, Otolaryngologist Head-Neck Surgeon, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0001-A
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Nasal Polyps
Keywords: Nasal polyps; Steroids; Prednisone; Nasal polypectomy; Blood loss, surgical
MeSH Terms: conditions — Nasal Polyps; Blood Loss, Surgical | interventions — Prednisone; Steroids; Adrenal Cortex Hormones; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone group (Experimental): Prednisone 50 mg daily for 10 days immediately pre-op
  Interventions: Drug: Oral Prednisone
- Placebo group (Placebo Comparator): Placebo pill for 10 days immediately pre-operative
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Oral Prednisone — Prednisone 50 mg once daily for 10 days pre-op
  Other Names: steroids; corticosteroids
  Arms: Prednisone group
Drug: Placebo comparator — Placebo pill identical to Prednisone 10 days once daily pre-op
  Other Names: sugar pill
  Arms: Placebo group

SUMMARY:
This study aims to determine if a short course of oral prednisone helps to improve the operative field and ease of surgery by minimizing bleeding during nasal polypectomy surgery.

DETAILED DESCRIPTION:
This study will be conducted as a double blinded randomized control trial and aims to recruit about 34 patients (17 patients per arm). Patients will be randomized to receive either prednisone 50 mg po x10 days or an identical looking placebo x10 days. Photographs of the polyps will be taken prior to the intervention, on the day of surgery and in the follow-up visit. Symptom survey (SNOT22) will also be administered at these same time points. Blood loss will be determined volumetrically from the suction canister and by using the Wormald Surgical field grading scale. Surgeons will also complete a survey postoperatively evaluating visibility, difficulty and ease of surgery. At 2 weeks, 1 month, 3 months and 6 months, patients will again fill out the Sino-nasal Outcome Test - 22 (SNOT-22) and the surgeon will do an endoscopic assessment by using the Peri-Operative Sinus Endoscopy (POSE) scoring system .

ELIGIBILITY:
Inclusion Criteria:

* All patients with severe obstructing nasal polyps scheduled for surgery.

Exclusion Criteria:

* Patient unable to tolerate side effects of prednisone
* Uncontrolled diabetes mellitus
* Hypertension
* Previous congestive heart failure
* Acute/chronic systemic infection
* History of hypersensitivity to prednisone
* History of cataracts or glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss. Wormald Surgical Field Grading Scale | Intraoperative
  This is an 11-point validated scale designed to provide a standardized method of documenting bleeding in endoscopic sinus surgery [Athanasiadis et al., 2007]. In addition blood loss during the surgery will be calculated from the suction canisters after accounting for the amount of irrigation used.
Visibility and easy of surgery | Immediate Postoperative period
  The surgeon will assess visibility and easy of surgery during the surgery and the technical difficulty of the surgery using two visual analogue scale questions.
Endoscopic assessment | 4 weeks, 3 months, 6 months
  The Peri-Operative Sinus Endoscopy (POSE) scoring system (total score) will be used to assess the condition of the patients' sinus cavities and the Lindholdt scale will be used to provide objective measures of polyp recurrence size based on the percent obstruction of the nasal cavity and obstruction based on anatomic location.

SECONDARY OUTCOMES:
Quality of life survey (SNOT22) | 2 weeks, 4 weeks, 3 months, 6 months post-op
  The Sino-nasal Outcome Test - 22 (SNOT-22) will be used as the main instrument to assess patients' disease specific symptoms. The total score from the SNOT-22 at 3 months follow-up will be the main outcome. The profile of symptom scores over the full follow-up period will be a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Witterick, MD FRCSC, Principal Investigator — University of Toronto Department of Otolaryngology-Head and Neck Surgery; Randy M Leung, BSc MD, Study Director — University of Toronto Department of Otolaryngology-Head and Neck Surgery
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, University of Toronto, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

REFERENCES:
- [Background] O'Driscoll BR, Kalra S, Wilson M, Pickering CA, Carroll KB, Woodcock AA. Double-blind trial of steroid tapering in acute asthma. Lancet. 1993 Feb 6;341(8841):324-7. doi: 10.1016/0140-6736(93)90134-3. PMID 8094111
- [Background] Hissaria P, Smith W, Wormald PJ, Taylor J, Vadas M, Gillis D, Kette F. Short course of systemic corticosteroids in sinonasal polyposis: a double-blind, randomized, placebo-controlled trial with evaluation of outcome measures. J Allergy Clin Immunol. 2006 Jul;118(1):128-33. doi: 10.1016/j.jaci.2006.03.012. Epub 2006 May 19. PMID 16815148
- [Background] Johansson L, Akerlund A, Holmberg K, Melen I, Stierna P, Bende M. Evaluation of methods for endoscopic staging of nasal polyposis. Acta Otolaryngol. 2000 Jan;120(1):72-6. doi: 10.1080/000164800760370873. PMID 10779190
- [Background] Sieskiewicz A, Olszewska E, Rogowski M, Grycz E. Preoperative corticosteroid oral therapy and intraoperative bleeding during functional endoscopic sinus surgery in patients with severe nasal polyposis: a preliminary investigation. Ann Otol Rhinol Laryngol. 2006 Jul;115(7):490-4. doi: 10.1177/000348940611500702. PMID 16900802
- [Background] Athanasiadis T, Beule A, Embate J, Steinmeier E, Field J, Wormald PJ. Standardized video-endoscopy and surgical field grading scale for endoscopic sinus surgery: a multi-centre study. Laryngoscope. 2008 Feb;118(2):314-9. doi: 10.1097/MLG.0b013e318157f764. PMID 17989575